CLINICAL TRIAL: NCT04486157
Title: A Phase 1, Open Label, Randomized, Single Dose, Two Treatment, Two Sequence, Two Period, Crossover Bioequivalence and Safety Study of IN-A012 and Akynzeo Capsules in Male and Female Healthy Korean Subjects
Brief Title: Bioequivalence and Safety Study of IN-A012 and Akynzeo Capsules in Male and Female Healthy Korean Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IN_FNP_101
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — netupitant, palosentron drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-A012 (Experimental): Intravenous administration of IN-A012
  Interventions: Drug: IN-A012
- Akynzeo capsules (Active Comparator): Single oral administration of Akynzeo capsules
  Interventions: Drug: Akynzeo 300Mg-0.5Mg Capsule

INTERVENTIONS:
Drug: IN-A012 — The subjects will be given IN-A012 by Intravenous infusion over 30 minutes.
  Arms: IN-A012
Drug: Akynzeo 300Mg-0.5Mg Capsule — The subjects will be administrated Akynzeo by Orally with water.
  Arms: Akynzeo capsules

SUMMARY:
The main purpose of this study is to demonstrate the bioequivalence between IN-A012 and Akynzeo capsules by pharmacokinetic(PK) evaluation

DETAILED DESCRIPTION:
[Pharmacokinetics Assessment]

* Primary Parameter

  - AUC0-t
* Secondary Parameters - Cmax, tmax

[Safety Assessment]

- Adverse events, vital signs, physical examination, 12-lead ECGs, and clinical laboratory tests

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged between 19-45
2. Body weight ≥ 50kg and in the range of ideal body weight ± 20%
3. Without congenital, or chronic diseases within recent 5 years
4. Subjects who are deemed eligible based on the screening tests
5. Subjects who received a full explanation of the study, understood the purpose and details of this study, characteristics of the investigational product, and expected adverse events, and voluntarily signed the informed consent form
6. Agree to use acceptable contraceptive methods from signing the informed consent to 3 weeks after the last dose of the investigational product
7. Able and willing to comply with study requirements including all scheduled inpatient and outpatient visits, clinical laboratory tests, and instructions.

Exclusion Criteria:

1. A subject with symptoms suspected of acute illness at the screening
2. A subject with clinically significant and active cardiovascular, respiratory, kidney, endocrine, hematological, gastrointestinal, central nervous system diseases, psychiatric disorders, or malignant tumors
3. A history of gastrointestinal disease
4. Known hypersensitivity to the active ingredient or excipients of investigational product or a history of clinically significant hypersensitivity
5. A history of drug abuse
6. Pregnant women or women who may be pregnant, and breastfeeding women
7. Subjects who are deemed inappropriate to participate in the study by the investigator for other reasons

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
AUC0-t of netupitant | pre-dose(0hour), 0.5, 1, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 , 120, 144, 168, 192, 216, and 240 hours post-dose
  Area under the plasma concentration versus time curve of netupitant

SECONDARY OUTCOMES:
Cmax of fosnetupitant, netupitant, netupitant metabolites and palonosetron | pre-dose(0hour), 0.5, 1, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 , 120, 144, 168, 192, 216, and 240 hours post-dose
  Peak Plasma Concentration of fosnetupitant, netupitant metabolites and palonosetron
tmax of fosnetupitant, netupitant, netupitant metabolites and palonosetron | pre-dose(0hour), 0.5, 1, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96 , 120, 144, 168, 192, 216, and 240 hours post-dose
  Time to reach maximum (peak) plasma concentration of fosnetupitant, netupitant, netupitant metabolites and palonosetron

CONTACTS AND LOCATIONS:
Overall Officials: Seunghoon Han, Principal Investigator — The Catholic University of Korea
Locations (1):
- Catholic Univ. of Seoul St. Mary's Hospital, Seoul, South Korea